CLINICAL TRIAL: NCT00396513
Title: Effect of Simvastatin and Metformin on Clinical, Endocrine, Metabolic and Endothelial Function of Women With Polycystic Ovary Syndrome: Prospective Randomised Trial
Brief Title: Simvastatin and Metformin Therapy in PCOS Women. Prospective Randomised Trial.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Poznan University of Medical Sciences (Other)
Collaborators: Yale University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1142/05
Record Dates: First submitted 2006-11-03; First posted 2006-11-07 (Estimated); Last update posted 2006-11-07 (Estimated); Status verified 2006-11

CONDITIONS: Polycystic Ovary Syndrome
Keywords: PCOS; Statin; Metformin; Testosterone; Menstrual cycle; Lipids
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Simvastatin; Metformin

INTERVENTIONS:
Drug: Simvastatin
Drug: Simvastatin and Metformin
Drug: Metformin

SUMMARY:
The purpose of this study is to compare effects of statins (simvastatin) and metformin on clinical (menstrual cycle, excessive hair, skin problems), endocrine (androgens), metabolic (lipids, markers of systemic inflammation), and endothelial function parameters in women with polycystic ovary syndrome (PCOS).

ELIGIBILITY:
Inclusion Criteria:

* PCO - ESHRE/ASRM criteria:oligomenorrhea (<8 spontaneus menses per year) and hyperandrogenism(hirsutism or acne) or hyperandrogenemia(testosterone > 70 ng/ml) normal prolactin, TSH, 17-OH progesterone no evidence of androgen producing malignancy, Cushing's syndrome or acromegaly age 18-40 reliable use of birth control pill for at least 3 months and no plans of pregnancy

Exclusion Criteria:

* elevated creatinine kinase above 2 times upper limit of normal or liver enzymes (transaminase) above 2 times of upper limit of normal use of any following medications: cyclosporine, fibrates niacin,antifungal agents, macrolide antibiotics use of oral contraceptives and other steroid hormones 3 months prior to the study

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 2005-09

PRIMARY OUTCOMES:
Serum testosterone

SECONDARY OUTCOMES:
regularity of menstrual cycle
serum lutropin
serum follitropin
serum lipids
serum DHEAS
serum SHBG
serum insulin

CONTACTS AND LOCATIONS:
Overall Officials: Leszek Pawelczyk, MD PhD, Principal Investigator — Poznan University of Medical Scienses; Antoni J Duleba, MD, Study Director — Yale University
Locations (1):
- Division of Infertility and Reproductive Endocrinology, Department of Gynecology and Obstetrics, Poznan, Poland

REFERENCES:
- [Derived] Xiong T, Fraison E, Kolibianaki E, Costello MF, Venetis C, Kostova EB. Statins for women with polycystic ovary syndrome not actively trying to conceive. Cochrane Database Syst Rev. 2023 Jul 18;7(7):CD008565. doi: 10.1002/14651858.CD008565.pub3. PMID 37462232
- [Derived] Banaszewska B, Pawelczyk L, Spaczynski RZ, Duleba AJ. Effects of simvastatin and metformin on polycystic ovary syndrome after six months of treatment. J Clin Endocrinol Metab. 2011 Nov;96(11):3493-501. doi: 10.1210/jc.2011-0501. Epub 2011 Aug 24. PMID 21865358
- [Derived] Banaszewska B, Pawelczyk L, Spaczynski RZ, Duleba AJ. Comparison of simvastatin and metformin in treatment of polycystic ovary syndrome: prospective randomized trial. J Clin Endocrinol Metab. 2009 Dec;94(12):4938-45. doi: 10.1210/jc.2009-1674. Epub 2009 Nov 4. PMID 19890022